CLINICAL TRIAL: NCT05584371
Title: Evaluation of the Safety and Tolerability of Exogenous Ketosis Induced by Free Beta-hydroxybutyrate.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: American Ketone LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UIE-4275-22-22-1
Record Dates: First submitted 2022-10-03; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Exogenous Ketosis
Keywords: Exogenous ketosis; Beta-hydroxybutyrate; Safety; Tolerability; Ketone bodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exogenous ketosis (Experimental): Intake of 10 grams of beta-hydroxybutyrate free of alcohol and salt.
  Interventions: Dietary Supplement: Free Beta-hydroxybutyrate

INTERVENTIONS:
Dietary Supplement: Free Beta-hydroxybutyrate — Participants will be asked to ingest 10 grams of beta-hydroxybutyrate, diluted in water and sweetened with Stevia, every morning between 9:00 and 11:00 for four weeks.
  Other Names: BetaFlow Ketone Concentrate

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of free beta-hydroxybutyrate induced ketosis in healthy individuals. The main question it aims to answer is:

* Is free beta-hydroxybutyrate safe and well tolerated by adults?

Participants will be asked to ingest 10 grams of beta-hydroxybutyrate, diluted in water and sweetened with Stevia, every morning between 9:00 and 11:00 for four weeks.

DETAILED DESCRIPTION:
Several ketogenic interventions have shown benefits in a wide variety of clinical scenarios. Ketosis can be induced in different ways: by 72 hours of fasting, with a carbohydrate-restricted diet and with supplements. For emergency situations, such as heart failure, the first two options are not an option for patients as they cannot wait 72 hours.

There are 3 safe supplements for inducing ketosis: ketone salts, ketone esters and medium-chain triglycerides. Even though they all raise the beta-hydroxybutyrate serum concentration, they significantly differ in safety profiles, drug vehicles, palatability and monetary costs. A biologically identical beta-hydroxybutyrate supplement with prompt onset of action and free of salt, alcohol and drug vehicles would be an adequate option in many clinical settings.

A gender and age-balanced adult sample will be recruited in order to evaluate the safety and tolerability of free beta-hydroxybutyrate. Participants will be asked to ingest 10 grams of beta-hydroxybutyrate, diluted in water and sweetened with Stevia, every morning between 9:00 and 11:00 for four weeks. Symptoms will be evaluated on a daily basis with a self-administered opened questionnaire. A venous blood gas analysis will be made at the beginning, 2 and 4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic adults who have not been diagnosed with chronic degenerative diseases or diseases that cause acid-base imbalances.
* Regarding women of childbearing age, it will only be recruited those who are using a method of contraception including oral contraception, contraceptive implant, contraceptive injection, intrauterine device (IUD) or patch.
* Adults without cognitive impairment that can compromise decision making.

Exclusion Criteria:

* Scheduled surgery during participation period.
* Adults on a ketogenic diet, carbohydrate-restricted diet or intermittent fasting.
* Women with a positive HCG serum or urine pregnancy test.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms | 4 weeks
  Frequency and severity of symptoms assessed by a self-administered questionnaire
Venous blood gas analysis | 4 weeks
  Analysis of pH, HCO3, CO2 and electrolytes to rule out disorders of acid-base balance

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Soto, PhD, MD., Principal Investigator — INCMNSZ
Locations (1):
- INCMNSZ, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Upon request to PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after publication
Access Criteria: Send email to adrian.sotom@incmnsz.mx

REFERENCES:
- [Background] Abe S, Ezaki O, Suzuki M. Medium-chain triglycerides (8:0 and 10:0) are promising nutrients for sarcopenia: a randomized controlled trial. Am J Clin Nutr. 2019 Sep 1;110(3):652-665. doi: 10.1093/ajcn/nqz138. PMID 31334544
- [Background] American Ketone. (n.d.). Therapeutic Ketosis = Potential for New Outcomes. Retrieved June 6, 2022, from https://americanketone.com
- [Background] Fortier M, Castellano CA, Croteau E, Langlois F, Bocti C, St-Pierre V, Vandenberghe C, Bernier M, Roy M, Descoteaux M, Whittingstall K, Lepage M, Turcotte EE, Fulop T, Cunnane SC. A ketogenic drink improves brain energy and some measures of cognition in mild cognitive impairment. Alzheimers Dement. 2019 May;15(5):625-634. doi: 10.1016/j.jalz.2018.12.017. Epub 2019 Apr 23. PMID 31027873
- [Background] Holland, A. M., Qazi, A. S., Beasley, K. N., & Bennett, H. R. (2019). Blood and cardiovascular health parameters after supplementing with ketone salts for six weeks. Journal of Insulin Resistance, 4(1), 7. https://doi.org/10.4102/jir.v4i1.47
- [Background] Nielsen R, Moller N, Gormsen LC, Tolbod LP, Hansson NH, Sorensen J, Harms HJ, Frokiaer J, Eiskjaer H, Jespersen NR, Mellemkjaer S, Lassen TR, Pryds K, Botker HE, Wiggers H. Cardiovascular Effects of Treatment With the Ketone Body 3-Hydroxybutyrate in Chronic Heart Failure Patients. Circulation. 2019 Apr 30;139(18):2129-2141. doi: 10.1161/CIRCULATIONAHA.118.036459. PMID 30884964
- [Background] Soto-Mota A, Norwitz NG, Clarke K. Why a d-beta-hydroxybutyrate monoester? Biochem Soc Trans. 2020 Feb 28;48(1):51-59. doi: 10.1042/BST20190240. PMID 32096539
- [Background] Soto-Mota A, Norwitz NG, Evans R, Clarke K, Barber TM. Exogenous ketosis in patients with type 2 diabetes: Safety, tolerability and effect on glycaemic control. Endocrinol Diabetes Metab. 2021 May 20;4(3):e00264. doi: 10.1002/edm2.264. eCollection 2021 Jul. PMID 34277987
- [Background] Soto-Mota A, Vansant H, Evans RD, Clarke K. Safety and tolerability of sustained exogenous ketosis using ketone monoester drinks for 28 days in healthy adults. Regul Toxicol Pharmacol. 2019 Dec;109:104506. doi: 10.1016/j.yrtph.2019.104506. Epub 2019 Oct 23. PMID 31655093
- [Background] St-Onge MP, Jones PJ. Physiological effects of medium-chain triglycerides: potential agents in the prevention of obesity. J Nutr. 2002 Mar;132(3):329-32. doi: 10.1093/jn/132.3.329. PMID 11880549
- [Background] Stubbs BJ, Cox PJ, Kirk T, Evans RD, Clarke K. Gastrointestinal Effects of Exogenous Ketone Drinks are Infrequent, Mild, and Vary According to Ketone Compound and Dose. Int J Sport Nutr Exerc Metab. 2019 Nov 1;29(6):596-603. doi: 10.1123/ijsnem.2019-0014. PMID 31034254